CLINICAL TRIAL: NCT03190538
Title: Nonalcoholic Steatohepatitis in Chinese Children: a Long Term Follow-up
Brief Title: Nonalcoholic Steatohepatitis in Chinese Children
Status: Recruiting | Type: Observational
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H&H_ChildNASH_01
Record Dates: First submitted 2017-06-10; First posted 2017-06-16 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver-biopsy will be collected and to be used as the diagnosis of NASH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There will be no specific intervention to these paediatric NASH patient

SUMMARY:
Nonalcoholic steatohepatitis (NASH) is now recognised as an increasing clinical problem in children. Steatosis without significant liver cell injury or fibrosis is the most common form of nonalcoholic fatty liver disease (NAFLD) in both adults and children. Studies in the adult population have variably suggested that steatosis is a benign nonprogressive condition and NASH is recognised as a potentially serious condition with significantly risk of morbidity and mortality.

A growing body of evidence suggests that children with NASH frequently show histopathological features that differ from those of adults. The prevalence of this pattern in a wide range of paediatric cases as well as other histopathological lesions and their relevance and prognostic significance in children with NAFLD remains to be determined. Thus the investigators would like to conduct a study of biopsies and clinical information to document the histological features of paediatric NAFLD, to explore the natural history of paediatric NAFLD, and to determine the frequency and prognostic value of these features.

ELIGIBILITY:
Inclusion Criteria:

* age 1-18 with biopsy-proven NAFLD
* Alcohol consumption less than 20g/day and 10g/day for boys and girls respectively

Exclusion Criteria:

* with viral hepatitis, e.g. HBV, HCV
* with a1-anti-trypsin disease
* with autoimmune hepatitis
* with Wilson disease
* with liver impaired by drugs

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with NAFLD who attended the Children's Liver Disease Center, 302 Hospital, Beijing, China will be identified and recruited. Participants met above inclusion and exclusion criteria will be invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Liver related death | Through study completion, an average of 1 year
  Whether the patients die from liver-related causes

SECONDARY OUTCOMES:
Complications of cirrhosis | Through study completion, an average of 1 year
  Whether the complication of cirrhosis i.e. ascites, hepatic encephalopathy, variceal bleeding occur during the follow-up
Liver biopsy | Through study completion, an average of 2 year
Liver transplant | Through study completion, an average of 1 year
  Whether the patients have liver transplant during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, PhD, Principal Investigator — Humanity and Health Medical Centre
Locations (1):
- Children's Liver Disease Center, 302 Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided